CLINICAL TRIAL: NCT05605951
Title: The Acute Optic Neuritis Network (ACON): a Non-interventional Prospective Multicenter Study on Diagnosis and Treatment of Acute Optic Neuritis
Brief Title: Acute Optic Neuritis Network: an International Study That Invesitages Subjects With a First-ever Episode of Acute Inflammation of the Optic Nerve
Acronym: ACON
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Experimental and Clinical Research Center, a cooperation between the Max Delbrück Center for Molecul (Other)
Responsible Party: Sponsor
Other Study IDs: ACON2022
Record Dates: First submitted 2022-10-23; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Demyelinating Diseases; Multiple Sclerosis; Neuromyelitis Optica Spectrum Disorder Attack; Myelin Oligodendrocyte Glycoprotein Antibody-associated Disease; Optic Neuritis
MeSH Terms: conditions — Demyelinating Diseases; Multiple Sclerosis; Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease; Optic Neuritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non-interventional study — observational study

SUMMARY:
The goal of this observational study is to longitudinally investigating subjects with inaugural acute optic neuritis (ON).

The main questions it aims to answer are:

* Does the time to corticosteroid treatment affect the visual outcome at 6 months in subjects with acute multiple sclerosis (MS)-, aquaporin 4-IgG positive (AQP4-IgG+) and myelin-oligodendrocyte-glycoprotein-IgG positive (MOG-IgG+) ON?
* How differ clinical, structural, and laboratory biomarkers in subjects with acute ON, including clinical isolated syndrome (CIS), MS-ON, AQP4-IgG+ON, MOG-IgG+ON and seronegative non-MS-ON? Participants will undergo
* clinical examination, including clinical history, neurovisual and neurological tests
* serum and cerebrospinal fluid examination
* optical coherence tomography (OCT)
* magnetic resonance imaging (MRI)
* assessment of depression, pain, quality of life through validated questionnaires Researchers will compare subjects with MS-ON, AQP4-IgG+ON, MOG-IgG+ON and other ON (CIS, seronegative non-MS-ON) to detect diagnostic and predictive markers for the disease course.

DETAILED DESCRIPTION:
The Acute Optic Neuritis Network (ACON) is a global cooperation of currently 26 academic centers longitudinally investigating subjects with inaugural acute optic neuritis (ON). ON often occurs at presentation of multiple sclerosis (MS), neuromyelitis optica spectrum disorders (NMOSD) and myelin-oligodendrocyte-glycoprotein (MOG) antibody-associated disease (MOGAD). The recommended treatment of high-dose corticosteroids for ON is based on a North-American study population, which did not address treatment timing, or antibody serostatus. The ACON study is primarily designed to investigate the effect of time to high-dose corticosteroid treatment on 6-month visual outcomes in ON.

All patients presenting within 30 days of inaugural ON will be enrolled. For primary analysis, patients will subsequently be assigned either into the MS-ON, aquaporin-4-IgG positive ON (AQP4-IgG+ON) or MOG-IgG positive ON (MOG-IgG+ON) group and then further sub-stratified according to the number of days from onset of visual loss to high-dose corticosteroids. The primary outcome measure will be high-contrast best-corrected visual acuity (HC-BCVA) at 6 months. Additionally, multimodal data will be collected in subjects with any ON (CIS-ON, MS-ON, AQP4-IgG+ON or MOG-IgG+ON and seronegative non-MS-ON), excluding infectious and granulomatous ON. Secondary outcomes include: optical coherence tomography (OCT) and magnetic resonance imaging (MRI) measurements, serum and cerebrospinal fluid (CSF) biomarkers (AQP4- and MOG-IgG levels; neurofilament; glial fibrillary protein), questionnaires (headache, visual function in daily routine, depression, and quality of life) at presentation, at 6- and 12-months follow-up. Data will be collected from 22 academic hospitals from Africa, Asia, the Middle East, Europe, North America, South America, Australia and Europe. Planned recruitment consists of 100 MS-ON, 50 AQP4-IgG+ON and 50 MOG-IgG+ON.

This prospective, multimodal data collection will assess the potential value of early high-dose corticosteroid treatment, investigate the interrelations between functional impairments and structural changes, and evaluate the diagnostic yield of laboratory biomarkers. This analysis has the ability to substantially improve treatment strategies and accuracy of diagnostic stratification in acute demyelinating ON.

ELIGIBILITY:
Inclusion Criteria:

* First-ever acute ON
* Onset of visual symptoms within maximum of 30 days
* Age ≥ 18 years
* Ability to give written informed consent
* Presence of written consent

Exclusion Criteria:

* MRI contraindication
* Prior demyelinating diagnosis
* Diagnosis of other forms of optic neuropathy (hereditary, granulomatous, infectious, infiltrative, toxic)
* Pregnancy at inclusion
* Relevant other diseases that conflict with study participation according to protocol
* Inability to cooperate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 300 patients with acute ON will be screened for study eligibility. We will include only inaugural ON patients. Subjects presenting for the first time with isolated ON or ON with additional demyelinating syndromes, e.g. myelitis or acute disseminated encephalomyelitis (ADEM) occurring within 30 days of the acute ON will be included. Patients with prior soft symptoms which can retrospectively be considered to be a demyelinating manifestation will be included, excluding patients with a prior demyelinating diagnosis. The prevalence of MS-, AQP4-IgG+ON and MOG-IgG+ON differs in each of the participating centers. For primary analysis, we collect data from subjects with MS-ON, AQP4-IgG+ON and MOG-IgG+ON. For secondary analysis, multimodal data will be collected in subjects with any demyelinating ON (CIS-ON, MS-ON, AQP4-IgG+ON or MOG-IgG+ON and seronegative non-MS-ON). We expect between 30-50% will be ineligible due to the rigorous exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
to investigate whether MS-ON, AQP4-IgG+ON and MOG-IgG+ON patients treated with early high-dose corticosteroids for visual loss have better visual outcomes and QoL than those with late treatment. | Six months follow-up
  visual acuity

SECONDARY OUTCOMES:
Visual and structural outcomes of acute ON in patients treated with high-dose corticosteroid-therapy versus plasmapheresis as first-line treatment. | Six months follow-up
  RNFL
Visual and structural outcomes of acute ON in patients treated with high-dose corticosteroid-therapy versus plasmapheresis as first-line treatment. | Six months follow-up
  MRI lesion score
Visual and structural outcomes of acute ON in patients treated with high-dose corticosteroid-therapy versus plasmapheresis as first-line treatment. | 12 months follow-up
  MRI lesion score
Visual and structural outcomes of MS-ON in patients treated with high-dose corticosteroid-therapy with oral prednisone taper vs. without taper as standard of care. | 12 months follow-up
  RNFL
Diagnostic and prognostic value of biomarker levels (NfL, GFAP) and associations with visual pathway damage (MRI- and OCT-based) in the acute stage and during follow-up. | Acute stage (onset)
  NfL (pg/ml)
Diagnostic and prognostic value of biomarker levels (NfL, GFAP) and associations with visual pathway damage (MRI- and OCT-based) in the acute stage and during follow-up. | Acute stage (onset)
  GFAP (pg/ml)
Diagnostic and prognostic value of biomarker levels (NfL, GFAP) and associations with visual pathway damage (MRI- and OCT-based) in the acute stage and during follow-up. | Six months follow-up
  NfL (pg/ml)
Diagnostic and prognostic value of biomarker levels (NfL, GFAP) and associations with visual pathway damage (MRI- and OCT-based) in the acute stage and during follow-up. | Six months follow-up
  GFAP (pg/ml)
Diagnostic and prognostic value of biomarker levels (NfL, GFAP) and associations with visual pathway damage (MRI- and OCT-based) in the acute stage and during follow-up. | 12 months follow-up
  NfL (pg/ml)
Diagnostic and prognostic value of biomarker levels (NfL, GFAP) and associations with visual pathway damage (MRI- and OCT-based) in the acute stage and during follow-up. | 12 months follow-up
  GFAP (pg/ml)
Characterization of MOG-IgG and AQP4-IgG levels and compartmentalisation (serum vs. CSF, using simultaneous paired samples) and associated risks for subsequent relapses in subjects with AQP4-IgG+ON and MOG-IgG+ON. | Acute stage (onset)
  MOG-IgG ratio
Characterization of MOG-IgG and AQP4-IgG levels and compartmentalisation (serum vs. CSF, using simultaneous paired samples) and associated risks for subsequent relapses in subjects with AQP4-IgG+ON and MOG-IgG+ON. | Acute stage (onset)
  AQP4-IgG ratio
Characterization of MOG-IgG and AQP4-IgG levels and compartmentalisation (serum vs. CSF, using simultaneous paired samples) and associated risks for subsequent relapses in subjects with AQP4-IgG+ON and MOG-IgG+ON. | Six months follow-up
  MOG-IgG IgG ratio
Characterization of MOG-IgG and AQP4-IgG levels and compartmentalisation (serum vs. CSF, using simultaneous paired samples) and associated risks for subsequent relapses in subjects with AQP4-IgG+ON and MOG-IgG+ON. | 12 months follow-up
  AQP4-IgG ratio
Diagnostic value of OCT markers (e.g. increased pRNFL) for diagnosis of MS, NMOSD, and MOGAD. | Acute stage (onset)
  pRNFL
Diagnostic value of OCT markers (e.g. increased pRNFL) for diagnosis of MS, NMOSD, and MOGAD. | Six months follow-up
  pRNFL
Prognostic value of OCT markers (e.g. increased pRNFL) for the visual outcome at 1-year follow-up. | 12 months follow-up
  pRNFL
Diagnostic value of OCT markers for a conversion from acute ON to clinically definite MS. | Acute stage (onset)
  OCT markers
Diagnostic value of OCT markers for a conversion from acute ON to clinically definite MS. | Six months follow-up
  OCT markers
Diagnostic value of OCT markers for a conversion from acute ON to clinically definite MS. | 12 months follow-up
  OCT markers
Diagnostic value of early clinical variables (i.e. visual loss and pain patterns). | Acute stage (onset)
  pain intensity
Diagnostic value of early clinical variables (i.e. visual loss and pain patterns). | Six months follow-up
  pain intensity
Diagnostic value of early clinical variables (i.e. visual loss and pain patterns). | 12 months follow-up
  pain intensity
Characterization of visual function in daily routine, visual QoL scores and incidence of depression at 1-year follow-up. | Six months follow-up
  NEI-VFQ-Score
Characterization of visual function in daily routine, visual QoL scores and incidence of depression at 1-year follow-up. | 12 months follow-up
  NEI-VFQ-Score
Characterization of visual function in daily routine, visual QoL scores and incidence of depression at 1-year follow-up. | Six months follow-up
  BDI-II Score
Characterization of visual function in daily routine, visual QoL scores and incidence of depression at 1-year follow-up. | 12 months follow-up
  BDI-II Score
Characterization of visual function in daily routine, visual QoL scores and incidence of depression at 1-year follow-up. | Six months follow-up
  EuroQol 5-Dimension EQ-5D-index
Characterization of visual function in daily routine, visual QoL scores and incidence of depression at 1-year follow-up. | 12 months follow-up
  EuroQol 5-Dimension EQ-5D-index

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Asseyer, Principal Investigator — Charite University, Berlin, Germany; Hadas Stiebel-Kalish, Principal Investigator — Rabin Medical Center, Tel Aviv
Locations (26):
- United States (3):
  - University of Colorado School of Medicine, Aurora, Colorado
  - Harvard Medical School, Boston, Massachusetts
  - Departments of Neurology and Ophthalmology, Mayo Clinic, Rochester, Minnesota
- Hospital Aleman, Buenos Aires, Argentina
- Department of Neurology, Concord Hospital, Faculty of Medicine and Health, Sydney, Australia
- University of Botswana, Gaborone, Botswana
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil
- Colombia (3):
  - Del Rosario University, Bogotá
  - Department of Ophthalmology, Oftlamo-Sanitas Eye Institute, School of Medicine, Fundación Universitaria Sanitas, Bogotá
  - Pontificia Universidad Javeriana, Bogotá
- Department of Neurology, Slagelse, Institute for Health Research, University of Southern Denmark, Odense, Denmark
- (MIRCEM) Lyon Civil Hospices, France, Lyon, France
- Germany (2):
  - Experimental and Clinical Research Center, Charité - Universitätsmedizin Berlin, Germany, Department of Neurology, Berlin
  - Institute for Clinical Neuroimmunology, LMU Clinic of Ludwig-Maximilians Universität in Munich, Munich
- Nitte University, Karnataka, Mangalore, India
- Israel (2):
  - Hadassah Hebrew University, Jerusalem
  - Sackler School of Medicine and Rabin Medical Center, Tel Aviv
- Italy (2):
  - University of Bologna, Bologna
  - University of Verona, Verona
- Fukushima Medical University School of Medicine, Fukushima, Japan
- National Cancer Center, Seúl University, Seoul, South Korea
- Spain (2):
  - University of Barcelona, Barcelona
  - Vall d'Hebron Barcelona Hospital Campus, Barcelona
- United Kingdom (2):
  - University Hospitals of Birmingham, Birmingham
  - Nuffield Department of Clinical Neurosciences, John Radcliffe Hospital, Oxford
- University Teaching Hospital in Lusaka, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analyzed during the current study are not publicly available but are available from the corresponding author upon reasonable request

REFERENCES:
- [Derived] Asseyer S, Asgari N, Bennett J, Bialer O, Blanco Y, Bosello F, Camos-Carreras A, Carnero Contentti E, Carta S, Chen J, Chien C, Chomba M, Dale RC, Dalmau J, Feldmann K, Flanagan EP, Froment Tilikete C, Garcia-Alfonso C, Havla J, Hellmann M, Kim HJ, Klyscz P, Konietschke F, La Morgia C, Lana-Peixoto M, Leite MI, Levin N, Levy M, Llufriu S, Lopez P, Lotan I, Lugaresi A, Marignier R, Mariotto S, Mollan SP, Ocampo C, Cosima Oertel F, Olszewska M, Palace J, Pandit L, Peralta Uribe JL, Pittock S, Ramanathan S, Rattanathamsakul N, Saiz A, Samadzadeh S, Sanchez-Dalmau B, Saylor D, Scheel M, Schmitz-Hubsch T, Shifa J, Siritho S, Sperber PS, Subramanian PS, Tiosano A, Vaknin-Dembinsky A, Mejia Vergara AJ, Wilf-Yarkoni A, Zarco LA, Zimmermann HG, Paul F, Stiebel-Kalish H. The Acute Optic Neuritis Network (ACON): Study protocol of a non-interventional prospective multicenter study on diagnosis and treatment of acute optic neuritis. Front Neurol. 2023 Feb 24;14:1102353. doi: 10.3389/fneur.2023.1102353. eCollection 2023. PMID 36908609